CLINICAL TRIAL: NCT05673213
Title: The Effects of Three-Stair Positioning Pillows Used for Preterm Infants on Physiological Parameters and Sleep-Wakefulness Status
Brief Title: Preterm Infants Physiological Parameters and Sleep-Wakefulness Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatma BOZDAG, Lecturer Doctor, Harran University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HRU-BOZDAG-002
Record Dates: First submitted 2023-01-01; First posted 2023-01-06 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Sleep

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine 15º head raised prone position (control group) (No Intervention): The infant was cared for, fed and treated by the primary nurse responsible for the infant between 08:30 and 08:55. No intervention was made to the preterm infant between 09:00-12:00 and the infant was allowed to rest. Preterm infants were followed for 3 hours (09:00-12:00) with routine 15º head raised prone position. Between these hours, the oxygen saturation and heart rate of the preterm infants in were counted by the researcher with a pulse oximeter device and recorded 18 times in 10 minutes. Sleep-wakefulness status was recorded by taking 15-second recordings with the Actigraphy measuring device.
- Three-stair positioning pillows group (Experimental): The infant was cared for, fed and treated by the primary nurse responsible for the infant between 08:30 and 08:55. No intervention was made to the preterm infant between 09:00-12:00 and the infant was allowed to rest. Preterm infants were followed for 3 hours (09:00-12:00) with three-stair positioning pillows. Between these hours, the oxygen saturation and heart rate of the preterm infants in were counted by the researcher with a pulse oximeter device and recorded 18 times in 10 minutes. Sleep-wakefulness status was recorded by taking 15-second recordings with the Actigraphy measuring device.
  Interventions: Other: Three-stair positioning pillows group

INTERVENTIONS:
Other: Three-stair positioning pillows group — The infant was cared for, fed and treated by the primary nurse responsible for the infant between 08:30 and 08:55. No intervention was made to the preterm infant between 09:00-12:00 and the infant was allowed to rest. Preterm infants were followed for 3 hours (09:00-12:00) with three-stair positioning pillows. Between these hours, the oxygen saturation and heart rate of the preterm infants in were counted by the researcher with a pulse oximeter device and recorded 18 times in 10 minutes. Sleep-wakefulness status was recorded by taking 15-second recordings with the Actigraphy measuring device.
  Arms: Three-stair positioning pillows group

SUMMARY:
This research was carried out between December 2021 and May 2022 as a randomized controlled experimental design. In the study, between 28-35 weeks of gestation preterm infants were divided into two groups as the experimental group (n=30) and the control group (n=30). The block randomization method was used to ensure that the infants were similar in terms of both weeks and weight due to the large interval between the weeks and to ensure the balance between the groups. Infants in the control group were followed in the routine prone position of the neonatal intensive care unit, while infants in the experimental group were followed in the prone position with three-stair positioning pillows.

DETAILED DESCRIPTION:
This research was carried a randomized controlled experimental design. The sample size in the study was 1.08, type 1 error was 5%, and statistical power was 95%, according to the power analysis performed by taking into account the Breathing frequency values of the groups in the study called "Effectiveness of Hammock Positioning in Reducing Pain and Improving Sleep-Wakefulness State in Preterm Infants". It was calculated as a total of 48 participants, 24 in each group (Ribas et al., 2019). Considering the possibility of losses, 30 preterm infants with TSPP (experimental) and 30 preterm infants who were not used (control) were included and the infants were randomly assigned to the groups. The block randomization method was used to ensure that the infants were similar in terms of both weeks and weight due to the large interval between the weeks and to ensure the balance between the groups. Infants were divided into 2 groups as 28-31 week gestation and 32-35 week gestation. 30 infants were randomly distributed to each gestational week group as experimental and control groups through a program available at http://www.randomizer.org. Families were informed by the researcher about the method of the study through face-to-face interviews, written and verbal consents were obtained, and the information about preterm infants and their families was recorded in the "Information Form". The actigraphy measuring device was connected to the computer and the device was installed by entering the parameters such as the name and surname of the infant to be treated and the time interval in which the recordings would be made. Data were collected from a single hall in the NICU. The noise level of the intensive care unit (NICU) was measured with the Uni-T UT353 Mini Decibelmeter Device and the average noise level of the hall where the data were collected was between 50-55 dB. The infant was cared for, fed and treated by the primary nurse responsible for the infant between 08:30 and 08:55. No intervention was made to the preterm infant between 09:00-12:00 and the infant was allowed to rest. Between these hours, the oxygen saturation and heart rate of the preterm infants in both groups were counted by the researcher with a pulse oximeter device and recorded 18 times in 10 minutes. Sleep-wakefulness status was recorded by taking 15-second recordings with the Actigraphy measuring device. Preterm infants in the experimental group were followed in the prone position with three-stair positioning pillows and the infants in the control group were followed in the routine 15º head raised prone position between the hours of the research follow-up. The study followed the CONSORT guideline for reporting randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Only being diagnosed as preterm as a result of the examination performed by the physician,
* Parent's willingness to participate in the research,
* The infant is between 28-35 weeks of gestation,
* Being in appropriate weight according to the week of gestation,
* Having a history of intubation and being extubated.

Exclusion Criteria:

* Surgical procedure has been applied,
* Diagnosed with sepsis,
* Congenital anomaly,
* Taking analgesics 4 hours before, which may affect sleep,
* Having hyperbilirubinemia,
* Having hypoglycemia,
* Presence of intracranial bleeding,
* Receiving any oxygen support (nasal O2, incubator O2, etc.),
* Intubated infants were not included in the study.

Ages: 28 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-05-28 (Actual)

PRIMARY OUTCOMES:
Sleep Status/minute | 3 hours
  Between 09:00-12:00
Wakefulness Status/minute | 3 hours
  Measurements were made with an actigraphy device between 09:00 and 12:00.
Physiological Parameters (oxygen saturation /%) | 3 hours
  Measurements were made with an actigraphy device between 09:00 and 12:00.
Physiological Parameters (heart rate/minute ) | 3 hours
  Between 09:00-12:00
Physiological Parameters (respiratory rate/minute ) | 3 hours
  Between 09:00-12:00

CONTACTS AND LOCATIONS:
Overall Officials: Fatma BOZDAĞ, Lecturer, Principal Investigator — Harran University
Locations (1):
- Harran University, Şanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No